CLINICAL TRIAL: NCT02274168
Title: Aid of Recording ICD Electrograms During Monomorphic Ventricular Tachycardia Ablation Procedures
Brief Title: Utility of ICD Electrograms During Ventricular Tachycardia Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Hospital de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIDEG-VTA
Record Dates: First submitted 2014-09-14; First posted 2014-10-24 (Estimated); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Sustained Monomorphic Ventricular Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional RF catheter ablation (Other): Conventional RF ablation will be performed without using ICD-EG information
  Interventions: Procedure: Conventional RF catheter ablation
- Investigational RF Catheter Ablation using ICD-EG information (Other): RF Catheter Ablation will be performed using ICD-EG information
  Interventions: Procedure: Investigational RF Catheter Ablation using ICD-EG information

INTERVENTIONS:
Procedure: Conventional RF catheter ablation — RF catheter ablation will be performed as usually done by each center. No ICD EGMs will be obtained and used during the ablation procedure (do not place the programming head over the ICD generator).
  Arms: Conventional RF catheter ablation
Procedure: Investigational RF Catheter Ablation using ICD-EG information — RF ablation procedure will be performed with the programming head over the ICD generator. ICD EGMs will be registered every time VT is induced and during ventricular pacing. ICD EGMs obtained during ablation procedure will be compared with the EGMs of the registered spontaneus VT and used to locate appropriate ablation sites.
  Arms: Investigational RF Catheter Ablation using ICD-EG information

SUMMARY:
With the increasing use of implantable cardioverter defibrillators (ICD) for primary prevention in patients with structural heart disease, an increasing number of patients are expected to develop their first episode of monomorphic ventricular tachycardia (VT) after an ICD is in place and the only documentation of the clinical arrhythmia will be the ICD electrogram (EG). The absence of a 12-lead ECG in patients with an ICD and sustained monomorphic VT represents a limitation when performing treatment with radiofrequency (RF) ablation. The analysis of ICD-EG during a RF ablation procedure is expected to provide a reference "model" of VT with clinical expression consisting of the electrical signal of the ICD during VT (which otherwise is not generally possible to obtain in ICD patients). This will allow for a more targeted approach to the substrate of the VT with clinical expression because: 1) if VT is induced by programmed stimulation, one can tell whether it is with clinical expression or not, and 2) if VT is not induced, ventricular pacing could be performed based on the comparative analysis of morphology and activation times of ICD-EG. These approaches will result in improved outcomes of the ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Clinical indication for RF catheter ablation
* Presence of an implanted ICD
* At least 1 episode of spontaneous sustained monomorphic VT documented with ICD electrogram
* Presence of structural heart disease
* Able to obtain signed informed consent and willing to comply with study activity requirements

Exclusion Criteria:

* It is anticipated that data can not be obtained during follow-up
* Unwilling or unable to provide informed consent
* Women who are or may potentially be pregnant
* Patients who are participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2011-04; Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients free of VT recurrence | 6 months

SECONDARY OUTCOMES:
Reduction in number of VT recurrence | 6 months
Reduction in the proportion of patients free of VT recurrence | 6 months
Reduction in the proportion of patients free of recurrence in patients in whom 12-lead ECG of the spontaneous VT is not available and in those in whom hemodinamically tolerated VT is not induced | 6 months and total follow-up
Improvement of spatial resolution of the ICD-EG after information from local ventricular endocardial acceleration is added | 6 months
  This outcome will be studied from the stored signal together with the ICD-EG on the device in the subgroup of patients with a device that allows to obtain this parameter. In the remaining patients, signals will be obtained noninvasively with a seismocardiogram using a highly sensitive accelerometer located in the sternal midline of the xiphoid process and simultaneously synchronized with the ECG.

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Almendral, MD, Study Director — HM hospitales
Locations (14):
- Spain (14):
  - Hospital General Universitario, Alicante
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Insular de Gran Canaria, Las Palmas
  - HM Hospitales, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Nuestra Señora de Valme, Seville
  - Hospital Virgen de la Salud, Toledo
  - Hospital Clínico Universitario, Valencia

REFERENCES:
- [Background] Yoshida K, Liu TY, Scott C, Hero A, Yokokawa M, Gupta S, Good E, Morady F, Bogun F. The value of defibrillator electrograms for recognition of clinical ventricular tachycardias and for pace mapping of post-infarction ventricular tachycardia. J Am Coll Cardiol. 2010 Sep 14;56(12):969-79. doi: 10.1016/j.jacc.2010.04.043. PMID 20828650
- [Background] Almendral J, Marchlinski F. Is it the same or a different ventricular tachycardia?: an additional use for defibrillator electrograms. J Am Coll Cardiol. 2010 Sep 14;56(12):980-2. doi: 10.1016/j.jacc.2010.03.081. No abstract available. PMID 20828651
- [Background] Almendral J, Atienza F, Everss E, Castilla L, Gonzalez-Torrecilla E, Ormaetxe J, Arenal A, Ortiz M, Sanroman-Junquera M, Mora-Jimenez I, Bellon JM, Rojo JL. Implantable defibrillator electrograms and origin of left ventricular impulses: an analysis of regionalization ability and visual spatial resolution. J Cardiovasc Electrophysiol. 2012 May;23(5):506-14. doi: 10.1111/j.1540-8167.2011.02233.x. Epub 2011 Dec 8. PMID 22151407